CLINICAL TRIAL: NCT00523705
Title: Escitalopram for Premenstrual Syndrome (PMS) in Teens: A Pilot Study
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Enrollment too slow.
Sponsor: University of Pennsylvania (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 805778; LXP-MD-123 (Forest Pharm) (Other: Forest Research Institute); LXP-MD-123 (Other: Forest Research Institute)
Record Dates: First submitted 2007-08-30; First posted 2007-08-31 (Estimated); Results first posted 2014-06-06 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2012-06

CONDITIONS: PMS
Keywords: premenstrual syndrome; PMS; PMDD; treatment; SSRI
MeSH Terms: conditions — Premenstrual Syndrome | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- escitalopram (Experimental): Escitalopram 10 mg tablets taken once daily. Dosing in the luteal phase of the menstrual cycle (estimated day 14 to day 2). Start at 10 mg/day (1 tablet) in the first treatment cycle. If unimproved, increase to 20 mg/day (2 tablets) in cycle 2 if not precluded by side effects.
  Interventions: Drug: escitalopram
- placebo (Placebo Comparator): Placebo tablets matched to drug.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: escitalopram — 10 mg tablets taken once daily. Dosing in the luteal phase of the menstrual cycle (estimated day 14 to day 2). Start at 10 mg/day (1 tablet) in the first treatment cycle. If unimproved, increase to 20 mg/day (2 tablets) in cycle 2 if not precluded by side effects.
  Other Names: Lexapro
  Arms: escitalopram
Other: placebo — Placebo tablets matched to drug
  Arms: placebo

SUMMARY:
The purpose of this pilot study is to determine the efficacy and safety of escitalopram administered premenstrually (day 14 through day 2 of the menstrual cycle) for severe PMS in young women ages 15-19 years.

DETAILED DESCRIPTION:
The medication in this study is a serotonin reuptake inhibitor (SSRI), a class that is considered the first-line treatment for severe PMS at this time. Although data indicate that young women who have PMS in their teen years report the same symptoms and symptom severity as adult women, clinical trials have not included this age group, and there is no information on the efficacy and safety of treatment with a serotonergic antidepressant for PMS in teens.

ELIGIBILITY:
Inclusion Criteria:

* Females 15-19 years of age
* Regular menstrual cycles of 22-35 days
* In general good health
* Medically approved birth control method if sexually active
* Evidence of ovulation
* Meeting all symptom criteria for PMS
* Signed informed consent
* Subjects under age 18 must also have signed parental consent

Exclusion Criteria:

* Current use of any treatment for PMS.
* Psychotropic or other medications that may compromise the study drug.
* Pregnancy, intending pregnancy or breast feeding.
* Not using a medically approved birth control method if sexually active.
* Significant medical or gynecological abnormalities.
* Irregular menses, any gynecologic disorder.
* Any severe or unstable medical illness.
* Any current major psychiatric diagnosis or any history of a major psychiatric diagnosis.
* Any current or history of alcohol abuse, drug abuse, suicide attempt, bi-polar disorder, psychosis or severe personality disorder.
* Use of triptans (Imitrex, Zomig, Frova, Maxalt, Axert, Amerge, Relpax).
* Use of medicines that include dextromethorphan such as Tylenol or Vicks cough medicines.
* Use of the pain medication meperidine.
* Use of any herbal product such as St John's Wort that may increase serotonin.
* Use of monoamine oxidase inhibitors (MAOIs), pimozide or citalopram hydrobromide.
* Drugs metabolized by CYP2D6 or a combination of CYP3A4 and CYP2D6 inhibitors.
* Hypersensitivity to escitalopram or citalopram.

Ages: 15 Years to 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2008-02; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Freeman, Principal Investigator — University of Pennsylvania
Locations (1):
- Dept OB/GYN, Mudd Professorship Suite, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Vichnin M, Freeman EW, Lin H, Hillman J, Bui S. Premenstrual syndrome (PMS) in adolescents: severity and impairment. J Pediatr Adolesc Gynecol. 2006 Dec;19(6):397-402. doi: 10.1016/j.jpag.2006.06.015. PMID 17174829

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period was from 01/25/08 to 07/07/09. The study was conducted in an academic research unit. 54 females signed consent for the study at visit 1. 43 were ineligible during the screen period and 11 were randomized to double-blind treatment.
Pre-assignment Details: During the screen period of 2 menstrual cycles, subjects rated daily symptom diaries to indicate the presence and severity of premenstrual symptoms. A total premenstrual score >80 in each cycle was required for randomization.
Groups:
- Sugar Pill: Placebo tablets matched to drug.
Period: Overall Study
Arm/Group | Escitalopram | Sugar Pill
Started | 7 | 4
Completed | 7 | 3 (1 withdrew due to no time)
Not Completed | 0 | 1
Not completed — No time for study. | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Escitalopram | Sugar Pill | Total
Number analyzed (Participants) | 7 | 4 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 4 | 11
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 17.6 (1.4) | 17.3 (1.3) | 17.4 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 4 | 11

OUTCOME MEASURES:

1. Primary Outcome: Subject Daily Symptom Rating Score.
Description: A daily diary with 17 symptoms of PMS rated on a 5-point scale to indicate none to very severe symptoms. Minimum score 0; maximum score 408.
Time Frame: baseline and 5 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Escitalopram | Sugar Pill
Number analyzed (Participants) | 7 | 4
units on a scale
  mean score at baseline | 155.6 (55.3) | 169 (59.1)
  mean score at endpoint (5 months) | 91.6 (54.2) | 121.3 (131.6)
Statistical Analysis 1: Comparison: Escitalopram vs Sugar Pill; Pilot data were examined at treatment endpoint for change from baseline. Statistical power was very low due to the small sample size; Test type: Superiority or Other; p = 0.467, Regression, Linear; Mean Difference (Final Values) = 3.57, Standard Error of Mean 4.86 — estimate of main effect of treatment in a linear mixed effects model

2. Secondary Outcome: Sheehan Disability Scale (SDS)
Time Frame: Throughout study
Population: Data not analyzed due to only 11 subjects.
Arm/Group | Escitalopram | Sugar Pill
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Patient Global Evaluation of Improvement (PGE)
Time Frame: Throughout treatment
Population: Not analyzed due to small number of subjects
Arm/Group | Escitalopram | Sugar Pill
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Subject Satisfaction Questionnaire
Time Frame: Study endpoint
Population: Not analyzed due to small number of subjects.
Arm/Group | Escitalopram | Sugar Pill
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 treatment months
Arm/Group | Escitalopram | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/4
Other Adverse Events (participants affected / at risk) | 5/7 | 0/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Escitalopram (N=7) | Sugar Pill (N=4)
fatigue (General disorders) | 3 (8) | 0 (0)
headache (Nervous system disorders) | 2 (2) | 0 (0)
nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
insomnia (General disorders) | 1 (1) | 0 (0)
breast tenderness (Reproductive system and breast disorders) | 1 (1) | 0 (0)
dizziness (Nervous system disorders) | 1 (1) | 0 (0)
other (General disorders) | 3 (6) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No